CLINICAL TRIAL: NCT04388631
Title: Detection Rate of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) in Male Genitourinary System and Its Impact on Male Reproductive Health: an Observational Clinical Study.
Brief Title: Detection Rate of SARS-CoV-2 in Male Genitourinary System and Its Impact on Male Reproductive Health.
Acronym: COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Jihong Liu, Principal Investigator, Clinical Professor, Tongji Hospital
Other Study IDs: 2020-S073
Record Dates: First submitted 2020-05-12; First posted 2020-05-14 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Coronavirus Disease 2019
Keywords: Coronavirus Disease 2019; Male reproductive health; Mental health
MeSH Terms: conditions — COVID-19; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — whole blood，serum，urine, prostate fluid, and semen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposed group: Male patient discharged with COVID-19
  Interventions: Other: Coronavirus Disease 2019
- Control group: Healthy male volunteers without COVID-19

INTERVENTIONS:
Other: Coronavirus Disease 2019 — male patients who have developed COVID-19
  Groups: Exposed group

SUMMARY:
This study will evaluate the changes in sexual function, reproductive function and mental health of male patients discharged from the hospital with COVID-19, and the impact of SARS-CoV-2 on male reproductive health and mental health compared with healthy people during the same period. In addition, men's semen examination reports before and after the new coronavirus pneumonia event will be collected and compared to assess the impact of the event on the quality of men's semen. Also, This study will test the SARS-CoV-2 nucleic acid of the urogenital system of male patients discharged with COVID-19 to provide evidence for the effect of the new coronavirus on the male reproductive system.

DETAILED DESCRIPTION:
This study will test SARS-CoV-2 nucleic acids in urine, prostate fluid, and semen of participants with COVID-19 at the first follow-up. All participants will be followed up for 1 year. During follow-up, International Index of Erectile Function-5 (IIEF-5), Quality Evaluation Questionnaire (QEQ), symptom list chart-90 (SCL-90) questionnaire evaluation and sexual function related examinations (including nocturnal penile tumescence, color duplex ultrasonography, etc. ) and fertility-related examinations (including sex hormones, semen routine examinations, etc.) will be performed to assess the changes in male sexual function, reproductive function and mental health of male patients discharged with COVID-19, and the impact of SARS-CoV-2 on male reproductive and mental health. In addition, collect male semen examination reports from April to December in 2017-2020 to evaluate the impact of new coronavirus pneumonia incidents on male semen quality.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥ 18, ≤ 60 years old;
2. Have a fixed sex partner and regular sex life;
3. No previous infectious diseases, chronic diseases, tumor history, and male sexual function and fertility diseases;
4. Normal erectile function, IIEF-5 score> 21 points;
5. Have complete clinical information and contact information；
6. Understand and sign the informed consent form.

Exclusion Criteria:

1. Hypertension, diabetes, coronary heart disease, hyperlipidemia and other chronic diseases；
2. Past history of endocrine diseases such as hypopituitarism, hypogonadism, abnormal thyroid function, etc;
3. Past history of mumps virus infection;
4. Past history of bladder cancer, prostate cancer, brain spine injury, testicular injury, pelvic fracture, urethral injury and history of surgical treatment;
5. Severe cardiovascular and cerebrovascular diseases, severe lung diseases, severe hepatitis;
6. Past psychological or mental illness;
7. Contact information not available.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — all participants are male
Study Population: male patients discharged with COVID-19 who have no previous sexual function and fertility related disease.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-05-10 (Estimated); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Sperm density | 3 months
  Sperm density will be obtained in the semen sample analysis using the World Health Organization (WHO) normal values based on the WHO 2010 reference limits.
Sperm activity | 3 months
  Sperm activity will be obtained in the semen sample analysis using the World Health Organization (WHO) normal values based on the WHO 2010 reference limits.
Erection hardness and duration | 3 months
  Erection hardness and duration will be evaluated during sleep by RigiscanHealth Organization (WHO) normal values based on the WHO 2010 reference limits.
IIEF-5/QEQ questionnaire score | 3 months
  IIEF-5/QEQ questionnaire score will be obtained by filling out the questionnaire every visit.
Detection rate of SARS-CoV-2 in male genitourinary system | 1 month
  Detection rate of SARS-CoV-2 in male genitourinary system will be evaluated by real time-polymerase chain reaction (RT-PCR).

SECONDARY OUTCOMES:
Semen volume | 3 months
  Sperm volume will be obtained in the semen sample analysis using the World Health Organization (WHO) normal values based on the WHO 2010 reference limits.
Sperm survival rate | 3 months
  Sperm survival rate will be obtained in the semen sample analysis using the World Health Organization (WHO) normal values based on the WHO 2010 reference limits.
Serum testosterone/luteinizing hormone (LH)/follicle stimulating hormone (FSH) level | 3 months
  The serum testosterone/LH/FSH levels will be tested in every visit.
SCL-90 questionnaire score | 3 months
  SCL-90 questionnaire score will be obtained using SCL-90 questionnaire.

OTHER OUTCOMES:
Height | 3 months
  Height will be measured at every visit
Weight | 3 months
  Weight will be measured at every visit
Clinical classification of COVID-19 | 1 month
  Clinical classification of COVID-19 will be determined according to the New Coronavirus Pneumonia Prevention and Control Program (7th edition) published by the National Health Commission of China

CONTACTS AND LOCATIONS:
Overall Officials: Jihong Liu, M.D, Principal Investigator — Departments of Urology, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, China
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measure will be available.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available with 6 months of study completion.
Access Criteria: Data access requests will be reviewed by the external independent review panel and Tongji hospital. Requester will be required to sign a Data Access Agreement.

REFERENCES:
- [Background] Hoffmann M, Kleine-Weber H, Schroeder S, Kruger N, Herrler T, Erichsen S, Schiergens TS, Herrler G, Wu NH, Nitsche A, Muller MA, Drosten C, Pohlmann S. SARS-CoV-2 Cell Entry Depends on ACE2 and TMPRSS2 and Is Blocked by a Clinically Proven Protease Inhibitor. Cell. 2020 Apr 16;181(2):271-280.e8. doi: 10.1016/j.cell.2020.02.052. Epub 2020 Mar 5. PMID 32142651
- [Background] Douglas GC, O'Bryan MK, Hedger MP, Lee DK, Yarski MA, Smith AI, Lew RA. The novel angiotensin-converting enzyme (ACE) homolog, ACE2, is selectively expressed by adult Leydig cells of the testis. Endocrinology. 2004 Oct;145(10):4703-11. doi: 10.1210/en.2004-0443. Epub 2004 Jul 1. PMID 15231706
- [Background] Xu J, Qi L, Chi X, Yang J, Wei X, Gong E, Peh S, Gu J. Orchitis: a complication of severe acute respiratory syndrome (SARS). Biol Reprod. 2006 Feb;74(2):410-6. doi: 10.1095/biolreprod.105.044776. Epub 2005 Oct 19. PMID 16237152
- [Background] Fraga-Silva RA, Costa-Fraga FP, Montecucco F, Sturny M, Faye Y, Mach F, Pelli G, Shenoy V, da Silva RF, Raizada MK, Santos RA, Stergiopulos N. Diminazene protects corpus cavernosum against hypercholesterolemia-induced injury. J Sex Med. 2015 Feb;12(2):289-302. doi: 10.1111/jsm.12757. Epub 2014 Nov 20. PMID 25411084